CLINICAL TRIAL: NCT02430090
Title: Comparison of Intratechal Low-Dose Levobupivacaine With Levobupivacaine-Fentanyl and Levobupivacaine-Sufentanil Combinations for Cesarean Section
Brief Title: Comparison of Intratechal Levobupivacaine and Adding With Sufetanil and Fentanyl in Ceserean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-099
Record Dates: First submitted 2015-04-20; First posted 2015-04-30 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2015-05

CONDITIONS: Anesthesia
Keywords: regionel anesthesia; levobupivacaine; ceserean section
MeSH Terms: interventions — Levobupivacaine; Fentanyl; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levobupivacaine (Experimental): Levobupivacaine, a local anesthetic agent, is indicated for the production of local or regional anesthesia or analgesia for surgery, for oral surgery procedures, for diagnostic and therapeutic procedures, and for obstetrical procedures.
  Injection Surgical anaesthesia
  Adult: Epidural block: 50-100 mg (10-20 ml) of a 0.5% solution or 75-150 mg (10-20 ml) of a 0.75% solution. Caesarean section: 75-150 mg (15-30 ml) of a 0.5% solution. Spinal block: 15 mg (3 ml) of a 0.5% solution. Max: 150 mg/dose; 400 mg/day. Injection Peripheral nerve block
  Read more: http://www.ndrugs.com/?s=levobupivacaine#ixzz3Xvp0iS5T
  Interventions: Drug: Levobupivacaine
- Levobupivacaine + fentanyl (Experimental): Fentanyl - Used for: Producing anesthesia for surgery and treating pain before, during, and after surgery.Fentanyl is a narcotic (opioid) analgesic. It works in the brain and nervous system to cause anesthesia and decrease pain.
  Indications:
  Adult: PO Breakthrough cancer pain As a loz: Initially, 200 mcg over 15 minutes for an episode of breakthrough pain; may repeat once after 15 minutes if needed. Not more than 4 unit doses/day. IV Adjunct to general anesth Patients w/ spontaneous resp: Initial: 50-200 mcg, w/ supplements of 50 mcg. Patients w/ assisted ventilation: Initial: 300-3,500 mcg (up to 50 mcg/kg), w/ supplements of 100-200 mcg depending on response.
  Read more: http://www.ndrugs.com/?s=fentanyl#ixzz3XvpAcULL
  Interventions: Drug: Fentanyl; Drug: Levobupivacaine
- Levobupivacaine + sufentanil (Experimental): Sufentanil is a synthetic opioid analgesic. Sufentanil exerts its principal pharmacologic effects on the central nervous system. Its primary actions of therapeutic value are analgesia and sedation.
  Maintenance: Additional doses of 0.5-10 mcg/kg may be given if needed. Max (total dose): 30 mcg/kg. Post-op pain Initial: 30-60 mcg. Additional doses of up to 25 mcg may be given at intervals of ≥1 hr if needed. Epidural Pain relief during labour and delivery W/ bupivacaine: 10-15 mcg w/ or w/o epinephrine. May repeat dose twice at intervals of ≥1 hr till delivery. Max (total dose): 30 mcg.
  Read more: http://www.ndrugs.com/?s=sufentanil#ixzz3XvqVyLzx
  Interventions: Drug: Sufentanil; Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — this used in intratechal area and for spinal anesthesia in ceserean section
  Other Names: chirocaine
  Arms: Levobupivacaine
Drug: Fentanyl — this used in intratechal area and for spinal anesthesia in ceserean section
  Arms: Levobupivacaine + fentanyl
Drug: Sufentanil — this used in intratechal area and for spinal anesthesia in ceserean section
  Other Names: sufenta
  Arms: Levobupivacaine + sufentanil
Drug: Levobupivacaine — this used in intratechal area and for spinal anesthesia in ceserean section
  Other Names: chirocaine
  Arms: Levobupivacaine + fentanyl
Drug: Levobupivacaine — this used in intratechal area and for spinal anesthesia in ceserean section
  Other Names: chirocaine
  Arms: Levobupivacaine + sufentanil

SUMMARY:
45 pregnant women undergoing cesarean section were enrolled in the study in november 2006 to march 2007. 2 ml of 0.5% levobupivacaine was added to 1 ml of saline in group I, 1 ml of 15 µcg of fentanyl in group II and 1 ml of 1,5 µcg sufentanil in group III by intratechal administration. Hemodynamic parameters, characteristics of sensory and motor blockade, peri-operative and postoperative visual analogue scale (VAS) pain scores, the time to the first analgesic requirement and adverse effects were recorded.

DETAILED DESCRIPTION:
45 pregnant women undergoing cesarean section were enrolled in the study in november 2006 to march 2007. Using CSE technique, 2 ml of 0.5% levobupivacaine was added to 1 ml of saline in group I, 1 ml of 15 µcg of fentanyl in group II and 1 ml of 1,5 µcg sufentanil in group III by intratechal administration. Hemodynamic parameters, characteristics of sensory and motor blockade, peri-operative and postoperative visual analogue scale (VAS) pain scores, the time to the first analgesic requirement and adverse effects were recorded.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with a single live fetus aged 18-45 years old and classified as ASA I, undergoing elective cesarean section, were included the study in november 2006 to march 2007

Exclusion Criteria:

* Multiple pregnancies,
* preterm labor,
* eclampsia,
* preeclampsia,
* concomitant diabetes mellitus,
* allergy to local anesthetics, fentanyl or sufentanil,
* contraindication for regional anesthesia were the exclusion criteria.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Müge Çakırca, Principal Investigator — Ankara Numune Training and Research hospital, Anesthesiology and Reanimation Clinic

REFERENCES:
- [Background] Stewart J, Kellett N, Castro D. The central nervous system and cardiovascular effects of levobupivacaine and ropivacaine in healthy volunteers. Anesth Analg. 2003 Aug;97(2):412-416. doi: 10.1213/01.ANE.0000069506.68137.F2. PMID 12873927
- [Background] Lee YY, Muchhal K, Chan CK. Levobupivacaine versus racemic bupivacaine in spinal anaesthesia for urological surgery. Anaesth Intensive Care. 2003 Dec;31(6):637-41. doi: 10.1177/0310057X0303100604. PMID 14719424
- [Background] Burke D, Kennedy S, Bannister J. Spinal anesthesia with 0.5% S(-)-bupivacaine for elective lower limb surgery. Reg Anesth Pain Med. 1999 Nov-Dec;24(6):519-23. doi: 10.1016/s1098-7339(99)90042-1. PMID 10588555

RESULTS

PARTICIPANT FLOW:
Groups:
- Levobupivacaine: Levobupivacaine, a local anesthetic agent, is indicated for the production of local or regional anesthesia or analgesia for surgery, for oral surgery procedures, for diagnostic and therapeutic procedures, and for obstetrical procedures.
  Injection Surgical anaesthesia
  Adult: Epidural block: 50-100 mg (10-20 ml) of a 0.5% solution or 75-150 mg (10-20 ml) of a 0.75% solution. Caesarean section: 75-150 mg (15-30 ml) of a 0.5% solution. Spinal block: 15 mg (3 ml) of a 0.5% solution. Max: 150 mg/dose; 400 mg/day. Injection Peripheral nerve block
  Read more: http://www.ndrugs.com/?s=levobupivacaine#ixzz3Xvp0iS5T
  Levobupivacaine: this used in intratechal area and for spinal anesthesia in ceserean section
- Levobupivacaine + Fentanyl: Fentanyl - Used for: Producing anesthesia for surgery and treating pain before, during, and after surgery.Fentanyl is a narcotic (opioid) analgesic. It works in the brain and nervous system to cause anesthesia and decrease pain.
  Indications:
  Adult: PO Breakthrough cancer pain As a loz: Initially, 200 mcg over 15 minutes for an episode of breakthrough pain; may repeat once after 15 minutes if needed. Not more than 4 unit doses/day. IV Adjunct to general anesth Patients w/ spontaneous resp: Initial: 50-200 mcg, w/ supplements of 50 mcg. Patients w/ assisted ventilation: Initial: 300-3,500 mcg (up to 50 mcg/kg), w/ supplements of 100-200 mcg depending on response.
  Read more: http://www.ndrugs.com/?s=fentanyl#ixzz3XvpAcULL
  Fentanyl: this used in intratechal area and for spinal anesthesia in ceserean section
  Levobupivacaine: this used in intratechal area and for spinal anesthesia in ceserean section
- Levobupivacaine + Sufentanil: Sufentanil is a synthetic opioid analgesic. Sufentanil exerts its principal pharmacologic effects on the central nervous system. Its primary actions of therapeutic value are analgesia and sedation.
  Maintenance: Additional doses of 0.5-10 mcg/kg may be given if needed. Max (total dose): 30 mcg/kg. Post-op pain Initial: 30-60 mcg. Additional doses of up to 25 mcg may be given at intervals of ≥1 hr if needed. Epidural Pain relief during labour and delivery W/ bupivacaine: 10-15 mcg w/ or w/o epinephrine. May repeat dose twice at intervals of ≥1 hr till delivery. Max (total dose): 30 mcg.
  Read more: http://www.ndrugs.com/?s=sufentanil#ixzz3XvqVyLzx
  Sufentanil: this used in intratechal area and for spinal anesthesia in ceserean section
  Levobupivacaine: this used in intratechal area and for spinal anesthesia in ceserean section
Period: Overall Study
Arm/Group | Levobupivacaine | Levobupivacaine + Fentanyl | Levobupivacaine + Sufentanil
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 45 female pregnant
Groups:
- Total: Total of all reporting groups
Arm/Group | Levobupivacaine | Levobupivacaine + Fentanyl | Levobupivacaine + Sufentanil | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (7.4) | 25.5 (5.2) | 27.4 (7.1) | 26.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 45
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 15 | 15 | 15 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: The frequency and the severity (ex) of the side effects including nausea and vomiting, hypotension, pruritus, and bradycardia were recorded.
Time Frame: Up to 4 months
Measure: Number; unit: participants
Groups:
- Levobupivacaine: 2 ml of 0.5% levobupivacaine was added to 1 ml of saline in group I by intrathecal administration
- Levobupivacaine + Fentanyl: 2 ml of 0.5% levobupivacaine was added to 1 ml of 15 µcg of fentanyl in group II by intrathecal administration
- Levobupivacaine + Sufentanil: 2 ml of 0.5% levobupivacaine was added to 1 ml of 1,5 µcg sufentanil in group III by intrathecal administration
Arm/Group | Levobupivacaine | Levobupivacaine + Fentanyl | Levobupivacaine + Sufentanil
Number analyzed (Participants) | 15 | 15 | 15
participants | 5 | 10 | 9

2. Secondary Outcome: Number of Participants With Pain Scores on the Visual Analog Scale
Description: Hemodynamic parameters, characteristics of sensory and motor blockade, peri-operative and postoperative visual analogue scale (VAS) pain scores, the time to the first analgesic requirement were recorded.
Time Frame: Up to 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Levobupivacaine | Levobupivacaine + Fentanyl | Levobupivacaine + Sufentanil
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 10/15 | 12/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levobupivacaine (N=15) | Levobupivacaine + Fentanyl (N=15) | Levobupivacaine + Sufentanil (N=15)
bradicardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) — <60 beat/minute
vomiting (General disorders) | 0 (0) | 2 (2) | 0 (0)
hypotension (General disorders) | 5 (5) | 10 (10) | 9 (9)
nausea (General disorders) | 1 (1) | 9 (9) | 8 (8)

LIMITATIONS AND CAVEATS:
A limitation of this study is that the baricity of the local anaesthetic could have been affected as the fentanyl and sufentanil were diluted within a mixture. Using these opiods in undiluted form in future studies would remove this limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No